CLINICAL TRIAL: NCT06099483
Title: Acute Effect of Motor Imagery Exercise Combined With Movement Observation on Brain Electrical Activity and Cardioventilatory Responses in Healthy Sedentary Individuals.
Brief Title: The Effect of Exercise on Brain Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, ebrar atak, Assistant Professor, Istanbul Gedik University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ebraratak1
Record Dates: First submitted 2023-10-16; First posted 2023-10-25 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary; EEG
Keywords: motor imagery; EEG; pulmonary rehabilitation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled double-blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- action observation and motor imegary (Active Comparator): The motor imagery and action observation group was asked to watch a previously recorded breathing exercise video and imagine it as if they were doing it themselves.
  Interventions: Other: Action observation and motor imagery
- Active Breathing Exercise Group (Active Comparator): Respiratory control, diaphragmatic breathing and thoracic expansion exercises were actively performed for 10 repetitions each.
  Interventions: Other: Active breathing exercise
- Control group (Active Comparator): Participants will remain in a sitting position throughout the entire experimental group application. Participants were prevented from making physical movements and were asked to keep their minds closed by closing their eyes and not thinking about anything.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Action observation and motor imagery — EEG recording was taken while watching a 10-minute video recording of specified breathing exercises and imagining the exercises.
  Arms: action observation and motor imegary
Other: Active breathing exercise — EEG recording was taken while the physiotherapist performed active breathing exercises for 10 minutes.
  Arms: Active Breathing Exercise Group
Other: Control group — EEG recording was taken while resting with eyes closed for 10 minutes.
  Arms: Control group

SUMMARY:
Concept of action simulation; It is an internal representation of motor programs that does not involve explicit movement. Motor imagery method (MI) or movement observation (HG) method are considered two separate action simulation methods that activate motor regions in the brain. Both methods remain a popular and effective tool for improving motor learning. Research has shown that clinicians working in rehabilitation settings are aware of the needs of patients, athletes, etc. are recommended as methods that participants can use to improve their motor skills.

Motor imagery training is a dynamic mental process in which a movement is mentally visualized without any visible movement or any voluntary motor muscle activation. Movement observation training is a method that involves internal, real-time motor simulation of movements in which the observer visually perceives movements performed by another. Mirror neurons, located primarily in the rostral part of the inferior parietal lobe and the ventral premotor cortex, are activated both when an action is physically performed and when the action is observed being performed by another person. Studies using neuroimaging techniques have provided support for this theory by showing that many areas known to be active during action simulation, such as the dorsal pre-motor cortex, supplementary motor area, superior parietal lobe, and intraparietal sulcus, are indeed active during both HG and MI. There is evidence in the literature that MI and HG also trigger sympathetic nervous system activation. There may be changes in respiration, heart rate and skin temperature, as well as an increase in electrodermal activity.

EEG is an inexpensive, noninvasive, and simple examination that can be used to evaluate neurophysiological functions by measuring electrical activity. Understanding the mechanism of beta rhythms is important because they are associated with conscious thinking, logical thinking, memory and problem solving, whereas suppression of beta waves contributes to depression and cognitive decline.

This study will investigate the effectiveness of exercising or watching or imagining exercise on brain functions.

DETAILED DESCRIPTION:
Participants in the study were divided into 3 groups. One group was shown breathing exercises and asked to imagine these exercises(Motor imagery and action observatin). The second group was made to do active exercises(The same exercises used in motor imagery and action observation were actively performed). The third group was not made to do anything. The exercises lasted 10 minutes. Watching and imagining the movement was also organized as a 10-minute program. That's why the control group was not allowed to do anything for 10 minutes. EEG recordings were taken during this 10-minute period in all three groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 18-40
* Not using an assistive device
* Having been using the same medications for the last 4 weeks
* No additional comorbid diseases of the orthopedic, neurological or cardiac system
* Getting 30 or more points from each of the Kinesthetic and Visual Imagination Questionnaire -20 (KGIA-20) visual imagination score and kinesthetic imagination score (The purpose of this criterion is to check that the patients who will be distributed to the cognitive rehabilitation group have sufficient imagination ability and to be able to do the exercises.)

Exclusion Criteria:

* Not agreeing to participate in the study
* Patients who have used oral corticosteroid drugs in the last 4 weeks
* Participants who cannot understand verbal instructions and are visually impaired
* Have currently participated in another clinical trial within the last 30 days that may affect the results of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Acute effect on brain electrical activity | up to 24 weeks
  Motor imagery exercise combined with action observation has an acute effect on brain electrical activity in healthy sedentary individuals.

SECONDARY OUTCOMES:
Acute effect on cardioventilatory responses | up to 24 weeks
  Motor imagery exercise combined with action observation has an acute effect on cardioventilatory responses in healthy sedentary individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrar Atak, PhD, Study Director — Istanbul Gedik University
Locations (1):
- Ebrar Atak, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atak E, Atac A. The Acute Effects of Motor Imagery Combined With Action Observation Breathing Exercise on Cardiorespiratory Responses, Brain Activity, and Cognition: A Randomized, Controlled Trial. Cardiovasc Ther. 2025 Feb 22;2025:6460951. doi: 10.1155/cdr/6460951. eCollection 2025. PMID 40026414